CLINICAL TRIAL: NCT03703011
Title: Accelerometers' Validity in Counting Number of Steps in the Elderly Subjects Before Discharge From Rehabilitation Units, Having Reached Their Maximal Walking Ability After Physiotherapy. Comparison of the Accuracy of 3 Accelerometer Positions: Wrist, Ankle, Hip
Brief Title: Accelerometers' Validity in Counting Number of Steps in the Elderly Subjects Before Discharge From Rehabilitation Units
Acronym: VAPODAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17004; 2018-A00348-47 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-04

CONDITIONS: Geriatrics
Keywords: geriatrics; discharge; Accelerometers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Subjects aged >70 years, hospitalized in the rehabilitation geriatric ward in the Paul Brousse hospital, France, able to walk 10 meters, ready to be discharged, and a Mini mental state examination ≥ 20/30
  Interventions: Device: Accelerometers positioned at the wrinkle, the hip, and the ankle

INTERVENTIONS:
Device: Accelerometers positioned at the wrinkle, the hip, and the ankle — Accelerometers are positioned at the wrinkle, the hip, and the ankle. The subject stands and walks 10 meters, followed up by a physiotherapist in the physiotherapy area. The accelerometers are triggered by a smartphone. The protocol is filmed (without the face), and 2 physicians will watch the film and count the steps blind to the results of the accelerometers (and blind to each-other steps counts)

SUMMARY:
Accelerometers enhance physical activity. Nevertheless, their validity (ability to accurately count steps) is not known in an elderly frail population ready for discharge from a rehabilitation unit. The objective was to assess accelerometers' validity for counting steps (10 meters), in comparison with the gold standard: steps counted by 2 physicians blind to accelerometers data, over a filmed 10-meter walk (minimal capacity to walk inside their own living place). The second objective was to evaluate the best position of the accelerometer: wrist, ankle, hip.

DETAILED DESCRIPTION:
Accelerometers enhance physical activity. Only one study assessed accelerometers' validly in an elderly robust population, over 100m walking distance. The accelerometers' validly was demonstrated especially for the ankle position (Floegel et al., 2017). The primary objective was to assess accelerometers validity for counting steps in an elderly frail population ready for discharge from a rehabilitation unit. The comparison gold standard was steps count by 2 physicians blind to accelerometers data, over a filmed 10-meter walk (minimal capacity to walk inside their own living place). The second objective was to evaluate the best position of the accelerometer: wrist, ankle, hip.

Investigators included prospectively subjects aged ≥ 70 years, hospitalized in the Paul Brousse geriatric rehabilitation ward, able to walk at least 10 meters (maximum functional recovery according to the physiotherapist opinion) and with a Mini mental state examination ≥ 20/30 (able to understand). All subjects gave written informed consent and the study was approved by the local ethics committee. The secondary objective was to evaluate the position of the accelerometer that give the most accurate step count: wrist, ankle, hip. The study took place in the Paul Brousse hospital in Villejuif in rehabilitations units. Falls during the protocol were considered as the only risk. To prevent this risk a physiotherapist walked behind the participants during the 10-meter walk. Demographic, clinical, physiological data were recorded and anonymized. In this monocentric non-randomized study, the number of participants to include was 120. Twenty participants were planned to be included each month during 6 months. Statistical analysis will be made by a T test to measure the difference between the gold standard and the count of the accelerometers. To eliminate measurement bias, Bland Altman analysis will be performed. Interclass correlation will be performed to measure the differences between accelerometers' positions. Logistic regressions will be done with measurement's variability determinants. In all analyses, the 2-sided α-level of 0.05 was used for significance testing.. All analysis will be performed using R statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Age> 70 years
* Patients able to walk 10 meters,
* Maximum functional recovery obtained according to the physiotherapist judgment and ready for discharge,
* Patients able to understand the instructions and to freely consent (Mini mental state examination ≥ 20/30 and score at the consent scale: UBACC≥ 12/20)
* Written consent
* Unprotected adult
* Covered by health insurance

Non inclusion Criteria:

* Impossibility to walk the required distance (severe dyspnea, post fall syndrome, blindness, ..)
* Patients participating in another interventional research.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Matching between number of steps measured by the accelerometers and the number of steps counted by the physicians visioning the film. | 3 days maximum (The 10-meter walk test is conducted within 3 days of signing the consent.)
  A step is counted when a foot touches the ground

SECONDARY OUTCOMES:
Matching between number of steps measured by the accelerometers worn on the ankle and the number of steps counted by the physicians visioning the film. | 3 days maximum (The 10-meter walk test is conducted within 3 days of signing the consent.)
  a step is counted when a foot touches the ground. Comparison between number of steps measured by the accelerometers worn on the ankle and the number of steps counted by the physicians visioning the film.
Matching between number of steps measured by the accelerometers worn on the wrist and the number of steps counted by the physicians visioning the film. | 3 days maximum (The 10-meter walk test is conducted within 3 days of signing the consent.)
  a step is counted when a foot touches the ground. Comparison between number of steps measured by the accelerometers worn on the wrist and the number of steps counted by the physicians visioning the film.
Best matching between the number of steps evaluated by the accelerometers and the the number of steps counted by the physicians visioning the film according to the accelerometers positions (hip, ankle, wrist). | 3 days maximum (The 10-meter walk test is conducted within 3 days of signing the consent.)
  a step is counted when a foot touches the ground. Comparison of the best matching between the number of steps evaluates by accelerometers worn on the hip, the ankle and the wrist and the number of steps counted by the physicians visioning the film.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle DURON, Md, PhD, Principal Investigator — APHP,Paul Brousse Hospital
Locations (1):
- Hopital Bicêtre - Geriatric Department, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No